CLINICAL TRIAL: NCT04175743
Title: Double-blinded, Placebo-controlled, Sequential Cohort, Multiple-Dose Escalation Study to Evaluate the Safety and Multiple Dose Pharmacokinetics of CT-044 HCl, a Reactive Species Decomposition Accelerant, in Healthy Human Volunteers
Brief Title: Double-blind, Placebo-control, Study to Evaluate the Safety and Pharmacokinetics of CT-044 HCl, in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lotus Clinical Research, LLC (Other)
Collaborators: CerSci Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CT044-002
Record Dates: First submitted 2019-11-06; First posted 2019-11-25 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Acute Pain; Pain, Acute; Surgery; Neuropathy
Keywords: Safety; Tolerability; Escalation; Pharmacokinetics; PK; CT-044 HCl; Ascending; Plasma; Surgical Pain; Acute Pain; Non-Opioid; Neuropathy; Chronic Neuropathy
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: The study is planned to have 3 dose levels (3 study cohorts); the actual dose level cohorts will be decided by the SRC after review of the data from each cohort that was successfully completed in the SAD study. Each dose cohort will include 8 subjects randomized to placebo (2 subjects) or active drug (6 subjects).
Who Masked: Participant, Investigator
Masking Description: Subjects will be assigned a randomization number prior to dosing on Day 1 in the order in which they are enrolled into the study to receive their allocated treatment according to a computer-generated randomization schedule prepared by the unblinded study statistician prior to the start of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 200 mg CT-044 HCl or Placebo (Experimental): 200 mg of CT-044 HCl administered every 8 hours vs placebo
  Interventions: Drug: CT-044 HCl
- 400 mg CT-044 HCl or Placebo (Experimental): 400 mg of CT-044 HCl administered every 8 hours vs placebo
  Interventions: Drug: CT-044 HCl
- 600 mg CT-044 HCl or Placebo (Experimental): 600 mg of CT-044 HCl administered every 8 hours vs placebo
  Interventions: Drug: CT-044 HCl

INTERVENTIONS:
Drug: CT-044 HCl — CT-044 HCl is a reactive species decomposition accelerant

SUMMARY:
This study will be conducted to assess safety, tolerability, and PK of CT-044 HCl in normal healthy volunteers, in a traditional sequential multiple ascending dose paradigm. The multiple-dose escalation is designed to mimic the manner in which the product (CT-044 HCl) would be used to manage ongoing pain in patients (i.e., multiple dosing).

DETAILED DESCRIPTION:
Subjects meeting all inclusion and exclusion criteria will be randomized to receive CT-044 HCl or placebo in three successive dose escalating cohorts of 8 subjects each (2 placebo and 6 active drug per dose level). Subjects will receive multiple oral CT-044 HCl doses for 7 days. Subjects will be monitored in-house for vital signs, physical examination, electrocardiogram (ECG), safety laboratory testing and documentation of adverse signs and symptoms. Serial blood and urine samples will be collected to evaluate CT-044 HCl levels in plasma and urine.

Eligible subjects will be admitted to the Clinical Trial Unit on the day prior to dosing (Day -1) and remain in house until Day 9 (discharge day). Subjects will return to the Clinical Trial Unit on an outpatient basis for follow-up (Day 13, ± 1 day).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index within the range 18.5 to 32.0 kg/m2 (inclusive).
* Healthy subjects as determined by medical history, physical examination including neurological examination, vital signs, electrocardiogram (ECG), and clinical laboratory tests.
* Negative tests for hepatitis B surface antigen, hepatitis C virus antibodies and human immunodeficiency virus (HIV-1 or HIV-2) antibody, and syphilis.
* Nonsmokers (use of any nicotine containing product) or ex-smokers (have ceased smoking for at least 3 months and do not use any drug for smoking cessation.
* Negative screen for alcohol and drugs of abuse.
* Women must not be of childbearing potential by reason of surgery or at least 1 year post-menopausal (i.e., 12 months without menstrual period), or menopause.
* Men must be infertile (at least 3-months post-vasectomy), or truly abstinent of heterosexual intercourse, or heterosexual partner is not of childbearing potential or must agree to use an effective method of contraception. Men must agree to not provide sperm donation during that same period.
* Able and willing to be available for the duration of the study.
* Willing and able to give written informed consent to participate.
* Able to understand and comply with protocol instructions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Maximum exposure level of CT-044 | 49 days
  Occurrence of maximum exposure level of Cmax of 80 μg/mL and/or AUC0-24 of 450 hr.μg/mL (corresponding to average values obtained at the NOAEL doses in males rat and dog) has been reached in ≥2 subjects in a cohort or if it is expected to be reached in the planned next cohort.
Plasma Pharmacokinetic Concentration of CT-044 | 32 Hours
  The PK data will be summarized by dose/cohort using appropriate statistics. Actual elapsed time from dosing will be used for the final plasma PK parameter calculations after database lock. Plasma PK samples collected every 8 hours for 32 hours.
Urine Pharmacokinetic Concentration of CT-044 | 24 Hours
  The urine PK concentration of CT-044 will use individual data points to determine the concentration of CT-044 in subjects urine. Urine PK samples collected every 8 hours for 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Lotus Clinical Resarch,LLC, Pasadena, California, United States

REFERENCES:
- [Derived] Squillace S, Salvemini D. Nitroxidative stress in pain and opioid-induced adverse effects: therapeutic opportunities. Pain. 2022 Feb 1;163(2):205-213. doi: 10.1097/j.pain.0000000000002347. No abstract available. PMID 34145168